CLINICAL TRIAL: NCT02243462
Title: Effectiveness of Pre-operative Warming in Prevention of Peri-operative Shivering
Brief Title: Preoperative Warming and Perioperative Shivering
Acronym: PWPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indus Hospital and Health Network (Other)
Responsible Party: Principal Investigator, Ali Asgher, Resident, Anesthesia, Indus Hospital and Health Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TIH-Anesth-001; IRD_IRB_2014_06_003 (Other: IRD IRB)
Record Dates: First submitted 2014-09-14; First posted 2014-09-18 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Forced Air Warming Effect on Hypothermia
Keywords: Shivering; Hypothermia; Postoperative; Temperature; Forced air warmer
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No pre-op warming (Other): No pre-warming in bay before surgery.
  Interventions: Other: No pre-op warming
- Pre-op forced air warming (Active Comparator): A forced air warmer device (WarmTouch Convective Warming System) will be used to pre-warm patients in holding bay before surgery
  Interventions: Device: Forced Air Warmer

INTERVENTIONS:
Device: Forced Air Warmer — A forced air warmer device will be used to pre-warm patients for 10 minutes in holding bay before surgery. Air warming device is an electrically powered control unit, hose, and inflatable "blanket". The control unit has an air filter and heater, which warms air entrained from the environment. The hose connects to a blanket.
  Other Names: WarmTouch Convective Warming System; Forced air warmer (FAW)
  Arms: Pre-op forced air warming
Other: No pre-op warming — No forced air warming of the patient prior to being taken in for surgery
  Arms: No pre-op warming

SUMMARY:
Shivering is one of the most commonly recognized problem associated with anesthesia, It is believed to be thermoregulatory in origin. Studies suggest that pre-warming the patient prior to the surgery can reduce the chances of hypothermia induced shivering during the post operative period.

Forced air warmers are the most frequently used active warming devices in the peri-operative setting. Currently, our hospital does not pre-warm patients but if our study shows that pre-warming reduces post-operative shivering, we will be able to make an evidence based decision to start this practice.

DETAILED DESCRIPTION:
Inadvertent peri-operative hypothermia (IPH) and shivering is one of the most commonly recognized problem during anesthesia which is believed to be thermoregulatory in origin. Although shivering is uncomfortable for most patients, it is unlikely that this relatively small increase in total body oxygen consumption in the average shivering patient is associated with increased peri-operative morbidity. It is common for patients to complain that their worst memory from the recovery room is the intense cold sensation and uncontrollable shivering. New guidelines recommend that patients core temperature has to be maintained at >36°C, postoperatively. Studies suggest that pre-warming the patient prior to the surgery can reduce the chances of hypothermia induced shivering during the post operative period.

Forced air warmers are the most frequently used active warming devices in the peri-operative setting. They are effective at preventing hypothermia induced shivering when used before induction of anesthesia, during anesthesia and surgery, and after emergence in the post-anesthesia care unit. Other methods such as warm fluids, opioids, blankets and warm light devices can be used but are less effective as compared to the forced air warming devices.

Currently, our hospital does not pre-warm patients but if our study shows that pre-warming reduces post-operative shivering, we will be able to make an evidence based decision to start this practice.

ELIGIBILITY:
Inclusion Criteria:

* All patients going under therapeutic laparoscopic surgery
* All patients between 15-70 years irrespective of their gender
* ASA 1-3 patients
* Those who have given informed consent

Exclusion Criteria:

* Any patient undergoing diagnostic laparoscopic surgery
* Patients below age of 15 yrs
* ASA 4 or higher patients
* Patients not giving informed consent

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
inadvertent shivering post surgery | upto 2-3 hours post-surgery
  number of patients who experience shivering in holding bay

CONTACTS AND LOCATIONS:
Overall Officials: Ali Asghar, MBBS, Principal Investigator — The Indus Hospital; Shahid Amin, Study Director — The Indus Hospital
Locations (1):
- The Indus Hospital, Karachi, Sindh, Pakistan